CLINICAL TRIAL: NCT04049032
Title: MUSC Women's Reproductive Behavioral Health Program for Opioid Use During Pregnancy
Brief Title: Perinatal Opioid Use
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00074655
Record Dates: First submitted 2019-08-01; First posted 2019-08-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Opioid Use; Pregnancy
Keywords: pregnancy; prescription opioids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- In-Person Participants: This group received perinatal OUD treatment in-person.
  Interventions: Behavioral: In-Person Perinatal OUD Treatment
- Telemedicine Participants: This group received perinatal OUD treatment via telemedicine.
  Interventions: Behavioral: Perinatal OUD Treatment via Telemedicine

INTERVENTIONS:
Behavioral: In-Person Perinatal OUD Treatment — Participants were seen weekly for four weeks, every two weeks for four weeks and monthly thereafter and provided relapse-prevention therapy and buprenorphine as part of standard of care.
  Groups: In-Person Participants
Behavioral: Perinatal OUD Treatment via Telemedicine — Participants were seen weekly for four weeks, every two weeks for four weeks and monthly thereafter and provided relapse-prevention therapy and buprenorphine as part of standard of care..
  Groups: Telemedicine Participants

SUMMARY:
To compare maternal and newborn outcomes among pregnant women with OUD receiving care via telemedicine versus in-person.

DETAILED DESCRIPTION:
Participants: Pregnant women with OUD.

Intervention: Participants were seen weekly for four weeks, every two weeks for four weeks and monthly thereafter and provided relapse-prevention therapy and buprenorphine.

Design: A cohort derived from a prospectively collected database including 98 women receiving perinatal OUD treatment in an obstetric practice by telemedicine or in-person and followed until 6-8 weeks postpartum from September, 2017 to December, 2018. Logistic regression with propensity score adjustment was applied to reduce group selection bias and control for potentially confounding variables.

Setting: Four outpatient obstetric practices in the southeast.

ELIGIBILITY:
Inclusion Criteria:

* Adult females, any race or ethnicity, age 18-45 years
* Currently pregnant
* Opioid Use Disorder (OUD)
* received in person or telemedicine treatment for OUD in their obstetrician's office

Exclusion Criteria:

* Not currently pregnant or receiving perinatal care
* Not in agreement with Patient-Physician Agreement

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: A cohort derived from a prospectively collected database including 94 women receiving perinatal OUD treatment in an obstetric practice by telemedicine or in-person and followed until 6-8 weeks postpartum from September, 2017 to December, 2018.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number of individuals retained in treatment | 6-8 weeks postpartum
  Uninterrupted addiction treatment during pregnancy through 6-8 weeks postpartum
Percent of infants born with Neonatal Abstinence Syndrome (NAS) | At Delivery
  Newborn withdrawal, also know as NAS gathered via electronic health record

SECONDARY OUTCOMES:
Positive urine drug screens | At delivery and 6-8 weeks postpartum
  Number of individuals with a positive urine drug screen
Length of newborn hospital stay and birth weight | Assessed up to 6 months following delivery
  Average number of days infant was in the hospital following delivery; weight of infant at birth

CONTACTS AND LOCATIONS:
Locations (1):
- The Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guille C, Simpson AN, Douglas E, Boyars L, Cristaldi K, McElligott J, Johnson D, Brady K. Treatment of Opioid Use Disorder in Pregnant Women via Telemedicine: A Nonrandomized Controlled Trial. JAMA Netw Open. 2020 Jan 3;3(1):e1920177. doi: 10.1001/jamanetworkopen.2019.20177. PMID 32003816